CLINICAL TRIAL: NCT02838693
Title: Assessing Progression to Type-2 Diabetes (APT-2D): A Prospective Cohort Study Expanded From BRITE-SPOT (Bio-bank and Registry for StratIfication and Targeted intErventions in the Spectrum Of Type 2 Diabetes)
Acronym: APT-2D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medicine (Other)
Collaborators: Janssen Pharmaceuticals (Industry); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor-Investigator, Medicine, Assistant Professor Sue-Anne Toh Ee Shiow, National University Hospital, Singapore
Organization: National University Hospital, Singapore (Other)
Other Study IDs: 28431754DIA4019
Record Dates: First submitted 2016-06-21; First posted 2016-07-20 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Pre-diabetes; Diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Storage of plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- APT-2D (Normoglycemic): 800 Normoglycemic
  Interventions: Procedure: Not applicable. This is an observational study.
- APT-2D (Pre-Diabetic): 1,500 Pre-Diabetic
  Interventions: Procedure: Not applicable. This is an observational study.

INTERVENTIONS:
Procedure: Not applicable. This is an observational study. — Not applicable. This is an observational study.

SUMMARY:
The Bio-bank and Registry for StratIfication and Targeted intErventions in the Spectrum Of Type 2 Diabetes (BRITE-SPOT) has been set up to prospectively collect clinical data and biologically relevant samples from individuals with, and at risk for type 2 diabetes (T2D), with the aim of delineating factors related to susceptibility, progression, complications and response to treatment. Expanded from BRITE-SPOT, Assessing the Progression to Type - 2 Diabetes (APT-2D) is a prospective cohort with a focus on non-diabetics (normoglycemic or prediabetic), to expand the sample size and depth of metabolic phenotyping in these upstream groups, with the more targeted aim of delineating factors related to insulin sensitivity versus secretion, that relate to progression to T2D.

DETAILED DESCRIPTION:
This is a prospective open cohort study.

The study will comprise the following periods:

Screening

• Complete screening checklist and informed consent form

Procedures.

* Following the screening visit, subjects are required to return to undergo the following:

  * Oral Glucose Tolerance Test (OGTT) to assess glucose tolerance and beta cell function
  * Frequently-Sampled Intravenous Glucose Tolerance test (FSIVGTT) to assess acute insulin response to glucose
  * Euglycemic Hyperinsulinemic Clamp (EHC) to obtain the insulin sensitivity index and assess insulin action
* The Disposition index (DI) that quantifies the relationship between insulin sensitivity and insulin secretion, will be determined through the results obtained during FSIVGTT and EHC to determine subject's risk for Type 2 diabetes.
* OGTT will be repeated every 6 months to assess for conversion to Type 2 Diabetes. Plasma C-peptide, and glucose will be measured at 7 time points during the OGTT for minimal model assessment of beta cell function
* FSIVGTT and EHC will be repeated within 3 months of conversion to Type 2 Diabetes, or at 3 years from recruitment, whichever comes sooner.

Normoglycemic Subjects: 800 Pre-Diabetic Subjects: 1500

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. At least 30 years old, and not older than 65 years
3. Overtly healthy males or females, as determined by medical history, physical examination and laboratory results
4. Not on any regular medications. Subjects using traditional medicine concomitantly will also be excluded in this study

Exclusion Criteria:

1. History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data
2. Known or ongoing psychiatric disorders within 3 years
3. Regularly use known drugs of abuse within 3 years
4. Women who are pregnant or lactating
5. Have donated blood of more than 500 mL within 4 weeks of study enrollment.
6. Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
7. Uncontrolled hypertension (blood pressure [BP] >160/100mmHg
8. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
9. Treatment with any investigational drug, or biological agent within one (1) month of screening or plans to enter into an investigational drug/ biological agent study during the duration of this study
10. Known allergy to insulin
11. History of bleeding diathesis or coagulopathy
12. Any of the following laboratory values at screening:

    * LDL > 190mg/dL (>4.9mmol/L)
    * TG > 500mg/dL (>5.6mmol/L)
    * Hba1C >= 6.5%
    * Fasting glucose >=126mg/dL(>=7mmol/L) or 2 hour post-prandial glucose >=200mg/dL (>=11.1mmol/L)
    * ALT > 3.0 x upper limit of normal
    * Estimated creatinine clearance <60 mL/min
13. Have any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study
14. Significant change in weight (+/- 5%) during the past month

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normoglycemic: 800 Pre-diabetics: 1,500
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2016-03; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes in beta-cell function in Asian populations with normal glucose tolerance and prediabetes over 3 years. | Data for each participant will be analysed upon completion all their OGTT visits
  Glucose & c-peptide laboratory results, from OGTT, will be used to assess glucose tolerance and beta cell function
Changes in insulin sensitivity in Asian populations with normal glucose tolerance and prediabetes over 3 years. Data will be presented at the end of 5.5years. | Data for each participant will be analysed upon completion of both of the FSIVGTT and EHC visits
  Disposition index assessed via glucose and insulin results from FSIVGTT and EHC.

SECONDARY OUTCOMES:
To discover and/or validate biomarkers that predict which subjects will progress from NGT to prediabetes and/or from prediabetes to diabetes. Data will be presented at the end of 5.5years. | All samples collected during the study will be consolidated at the end of 5.5years or upon study completion, whichever that comes first, and analysed in one single batch to ensure consistency of the data
  Biomarker panel will be conducted through testing of plasma and serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sue-Anne Toh, MBBChir, MSc, MA, Principal Investigator — mdcsates@nus.edu.sg
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Tai ES, Goh SY, Lee JJ, Wong MS, Heng D, Hughes K, Chew SK, Cutter J, Chew W, Gu K, Chia KS, Tan CE. Lowering the criterion for impaired fasting glucose: impact on disease prevalence and associated risk of diabetes and ischemic heart disease. Diabetes Care. 2004 Jul;27(7):1728-34. doi: 10.2337/diacare.27.7.1728. PMID 15220254
- [Background] Bergman RN, Phillips LS, Cobelli C. Physiologic evaluation of factors controlling glucose tolerance in man: measurement of insulin sensitivity and beta-cell glucose sensitivity from the response to intravenous glucose. J Clin Invest. 1981 Dec;68(6):1456-67. doi: 10.1172/jci110398. PMID 7033284
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Chen M, Porte D Jr. The effect of rate and dose of glucose infusion on the acute insulin response in man. J Clin Endocrinol Metab. 1976 Jun;42(6):1168-75. doi: 10.1210/jcem-42-6-1168. PMID 932179
- [Background] Dalla Man C, Campioni M, Polonsky KS, Basu R, Rizza RA, Toffolo G, Cobelli C. Two-hour seven-sample oral glucose tolerance test and meal protocol: minimal model assessment of beta-cell responsivity and insulin sensitivity in nondiabetic individuals. Diabetes. 2005 Nov;54(11):3265-73. doi: 10.2337/diabetes.54.11.3265. PMID 16249454
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Tan CE, Emmanuel SC, Tan BY, Jacob E. Prevalence of diabetes and ethnic differences in cardiovascular risk factors. The 1992 Singapore National Health Survey. Diabetes Care. 1999 Feb;22(2):241-7. doi: 10.2337/diacare.22.2.241. PMID 10333940
- [Background] Jin W, Patti ME. Genetic determinants and molecular pathways in the pathogenesis of Type 2 diabetes. Clin Sci (Lond). 2009 Jan;116(2):99-111. doi: 10.1042/CS20080090. PMID 19076063
- [Background] Levy J, Atkinson AB, Bell PM, McCance DR, Hadden DR. Beta-cell deterioration determines the onset and rate of progression of secondary dietary failure in type 2 diabetes mellitus: the 10-year follow-up of the Belfast Diet Study. Diabet Med. 1998 Apr;15(4):290-6. doi: 10.1002/(SICI)1096-9136(199804)15:43.0.CO;2-M. PMID 9585393
- [Background] Bagust A, Beale S. Deteriorating beta-cell function in type 2 diabetes: a long-term model. QJM. 2003 Apr;96(4):281-8. doi: 10.1093/qjmed/hcg040. PMID 12651972
- [Background] Turner R, Stratton I, Horton V, Manley S, Zimmet P, Mackay IR, Shattock M, Bottazzo GF, Holman R. UKPDS 25: autoantibodies to islet-cell cytoplasm and glutamic acid decarboxylase for prediction of insulin requirement in type 2 diabetes. UK Prospective Diabetes Study Group. Lancet. 1997 Nov 1;350(9087):1288-93. doi: 10.1016/s0140-6736(97)03062-6. PMID 9357409
- [Background] Matthews DR, Cull CA, Stratton IM, Holman RR, Turner RC. UKPDS 26: Sulphonylurea failure in non-insulin-dependent diabetic patients over six years. UK Prospective Diabetes Study (UKPDS) Group. Diabet Med. 1998 Apr;15(4):297-303. doi: 10.1002/(SICI)1096-9136(199804)15:43.0.CO;2-W. PMID 9585394
- [Background] Donnan PT, MacDonald TM, Morris AD. Adherence to prescribed oral hypoglycaemic medication in a population of patients with Type 2 diabetes: a retrospective cohort study. Diabet Med. 2002 Apr;19(4):279-84. doi: 10.1046/j.1464-5491.2002.00689.x. PMID 11942998
- [Background] Ringborg A, Lindgren P, Yin DD, Martinell M, Stalhammar J. Time to insulin treatment and factors associated with insulin prescription in Swedish patients with type 2 diabetes. Diabetes Metab. 2010 Jun;36(3):198-203. doi: 10.1016/j.diabet.2009.11.006. Epub 2010 Mar 28. PMID 20347376
- [Background] Cook MN, Girman CJ, Stein PP, Alexander CM, Holman RR. Glycemic control continues to deteriorate after sulfonylureas are added to metformin among patients with type 2 diabetes. Diabetes Care. 2005 May;28(5):995-1000. doi: 10.2337/diacare.28.5.995. PMID 15855556
- [Background] Zhou K, Donnelly LA, Morris AD, Franks PW, Jennison C, Palmer CN, Pearson ER. Clinical and genetic determinants of progression of type 2 diabetes: a DIRECT study. Diabetes Care. 2014;37(3):718-724. doi: 10.2337/dc13-1995. Epub 2013 Nov 1. PMID 24186880
- [Background] Kola I, Landis J. Can the pharmaceutical industry reduce attrition rates? Nat Rev Drug Discov. 2004 Aug;3(8):711-5. doi: 10.1038/nrd1470. No abstract available. PMID 15286737
- [Background] Riese DJ 2nd, Settleman J, Neary K, DiMaio D. Bovine papillomavirus E2 repressor mutant displays a high-copy-number phenotype and enhanced transforming activity. J Virol. 1990 Feb;64(2):944-9. doi: 10.1128/JVI.64.2.944-949.1990. PMID 2153255
- [Background] Paul SM, Mytelka DS, Dunwiddie CT, Persinger CC, Munos BH, Lindborg SR, Schacht AL. How to improve R&D productivity: the pharmaceutical industry's grand challenge. Nat Rev Drug Discov. 2010 Mar;9(3):203-14. doi: 10.1038/nrd3078. Epub 2010 Feb 19. PMID 20168317
- [Derived] Tsai MH, Goh CE, Lee MH, Seah F, Lim M, Febriana E, Fu J, Yip JK, Preshaw P, Toh SES. Associations between perceived stress and glycemic measures: gender and age as moderators. BMJ Open Diabetes Res Care. 2025 Nov 4;13(6):e005368. doi: 10.1136/bmjdrc-2025-005368. PMID 41192939